CLINICAL TRIAL: NCT06031272
Title: A Phase I, Randomized, Placebo-Controlled Study of the Safety, Antiviral & Immunomodulatory Activity of Broadly Neutralizing Antibodies 3BNC117-LS-J and 10-1074-LS-J in Combination in ART-treated Adults in Sub-Saharan Africa Living With HIV During a Monitored Analytical Treatment Interruption
Brief Title: Pausing Antiretroviral Treatment Under Structured Evaluation
Acronym: PAUSE
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5416; UM1AI068636 (NIH); HVTN 806 (Other: HIV Vaccine Trials Network (HVTN)); HPTN 108 (Other: HIV Prevention Trials Network (HPTN))
Record Dates: First submitted 2023-08-14; First posted 2023-09-11 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-01

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: 30 mg/kg 3BNC117-LS-J + 10 mg/kg 10-1074-LS-J (Experimental): Participants will receive 30 mg/kg 3BNC117-LS-J and 10 mg/kg 10-1074-LS-J, administered as two intravenous (IV) infusions at Step 1 entry (Day 0). Participants will discontinue ART on Day 2.
  Interventions: Drug: 3BNC117-LS-J; Drug: 10-1074-LS-J
- Arm B: Placebo (Placebo Comparator): Participants will receive dose-volume equivalent placebo IV infusions for both 3BNC117-LS-J and 10-1074-LS-J at Step 1 entry (Day 0). Participants will discontinue ART on Day 2.
  Interventions: Drug: Placebo for 3BNC117-LS-J; Drug: Placebo for 10-1074-LS-J

INTERVENTIONS:
Drug: 3BNC117-LS-J — Administered by intravenous (IV) infusion
  Arms: Arm A: 30 mg/kg 3BNC117-LS-J + 10 mg/kg 10-1074-LS-J
Drug: 10-1074-LS-J — Administered by intravenous (IV) infusion
  Arms: Arm A: 30 mg/kg 3BNC117-LS-J + 10 mg/kg 10-1074-LS-J
Drug: Placebo for 3BNC117-LS-J — Administered by intravenous (IV) infusion
  Arms: Arm B: Placebo
Drug: Placebo for 10-1074-LS-J — Administered by intravenous (IV) infusion
  Arms: Arm B: Placebo

SUMMARY:
The main purpose of this study is to see if it is safe to give the study antibodies (3BNC117-LS-J and 10-1074-LS-J) by intravenous infusion to people with HIV (PWH), and to see if they cause any side effects. In addition, to see how the study antibodies affect the level of HIV in the blood when participants are not taking regular HIV treatment for an extended period. This extended period of not taking regular HIV treatment is called an analytical treatment interruption (ATI).

ELIGIBILITY:
Inclusion Criteria:

Step 1:

* Ability and willingness of participant to provide informed consent.
* HIV-1 infection, documented by:

  * Any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry AND
  * Confirmed by one of the following:

    * A second antibody test from different manufacturers or based on different principles and epitopes (combination antigen-antibody-based rapid tests may be used)
    * HIV-1 antigen, or
    * Plasma HIV-1 RNA viral load, or
    * A licensed Western blot [NOTE: The term "licensed" refers to a U.S. FDA-approved kit.]
* On stable suppressive ART for at least 96 weeks prior to study entry. [NOTE: ART interruptions of up to 7 days occurring ≥90 days prior to study entry are acceptable. Within- and between-class changes in ART within the year prior to study entry are acceptable.]
* Plasma HIV-1 RNA levels of <50 copies/mL for at least 96 weeks prior to study entry at any licensed local laboratory or Network-approved non-US laboratory that is VQA certified.

[NOTE: Two "blips" (i.e., plasma HIV-1 RNA >50 and <400 copies/mL) are allowed if each blip is preceded and followed by values <50 copies/mL. At least one viral load measurement in greater than 56 days and within 48 weeks prior to the entry visit and another viral load within 56 days prior to the entry visit must be available for review. ]

* CD4+ cell count >450 cells/µL obtained within 56 days prior to study entry at any Network-approved non-US laboratory that is IQA certified.
* The following laboratory values obtained within 56 days prior to study entry by any Network-approved non-US laboratory that is EQA certified:

  * Absolute neutrophil count (ANC) ≥750/mm3
  * Hemoglobin ≥10 g/dL for participants who were assigned female sex at birth, ≥11.0 g/dL for participants who were assigned male sex at birth
  * Platelet count ≥100,000/mm3
  * Estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73m2 as calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) equation
  * ALT <2.5 times the institutional upper limit of normal
  * Direct bilirubin within the institutional range of normal
* For participants who can become pregnant (i.e., participants assigned female sex at birth who have not been post-menopausal for at least 24 consecutive months, who have had menses within the preceding 24 months, or who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy), negative serum or urine pregnancy test within 24 hours prior to Step 1 entry (Day 0) by a Network-approved non-US laboratory that is EQA certified. [NOTE: Participant-reported history is acceptable documentation of hysterectomy and bilateral oophorectomy, tubal ligation, tubal micro-inserts.]
* Participants who can become pregnant must agree to use two methods of contraception, one of which must be from the highly effective methods for contraception listed below. Barrier methods of contraception are permitted for the second method of contraception. Contraception must be used from 10 days prior to study entry and participants must agree to use contraception for 36 weeks after receiving study treatment, and until ART is reinitiated and viral suppression is achieved. Acceptable methods of contraception include:

  * Contraceptive subdermal implant
  * Intrauterine device or intrauterine system
  * Combined estrogen and progestogen oral contraceptive
  * Injectable progestogen
  * Contraceptive vaginal ring
  * Percutaneous contraceptive patches
  * Partner sterilization with documentation of azoospermia prior to the participant's entry into the study, and this partner is the sole partner for that participant. The documentation of partner sterility can come from the site personnel's review of medical records, medical examination and/or semen analysis, or medical history interview provided by the participant or the partner. Self-reported documentation of reproductive potential should be entered in the source documents.
* Participants who can impregnate (i.e., individuals assigned male sex at birth who have not undergone a sterilizing procedure) a partner and who are engaging in sexual activity that could lead to pregnancy must agree to use condoms from 10 days prior to study entry and for 36 weeks after receiving study treatment to avoid impregnating a partner.
* Willingness to use barrier protection (i.e., external or internal) for all sexual activity during ATI and until viral suppression is achieved after re-starting ART.
* Willingness to not participate in other research studies of investigational drugs while on this study.
* Willingness to provide a specimen for a genetic test (HLA Typing).

Step 2:

* Participant who has completed Step 1, including receipt of both bNAb infusions, and has not met ART restart criteria described in the protocol at any time during Step 1.
* Willingness to continue ATI and be monitored.

Step 3:

* Meeting one or more ART restart criteria described in the protocol OR
* Despite completing 72 weeks of ATI without meeting one or more ART restart criteria, participant declines participation in A5385, or is unable to enter A5385.

Exclusion Criteria:

Step 1:

* History of any AIDS-defining illness prior to study entry. [NOTE: History of treated and resolved pulmonary TB will not be exclusionary.]
* Known nadir CD4+ cell count <200 cells/µL. [NOTE: If laboratory reports or clinical notes are not available, then participant recall is acceptable for nadir CD4 T-cell count.]
* Any clinically significant acute or chronic medical condition (such as autoimmune diseases or active tuberculosis), other than HIV infection, that in the opinion of the investigator would preclude participation.
* Any history of an HIV-associated malignancy, including Kaposi's sarcoma, or any type of lymphoma or virus-associated cancers.
* History of Progressive Multifocal Leukoencephalopathy (PML).
* Active or recent non-HIV-associated malignancy requiring systemic chemotherapy or surgery within 36 months prior to study entry or for whom such therapies are expected in the subsequent 12 months. [NOTE: Minor surgical removal of localized skin cancers (squamous cell carcinoma, basal cell carcinoma) is not exclusionary.]
* Receipt of an NNRTI within 30 days prior to study entry.
* Receipt of cabotegravir-LA IM, rilpivirine-LA IM, or other long-acting ARVs within 24 months prior to study entry.
* Receipt of any standard-of-care (SOC) vaccines within 7 days prior to study entry.
* Known resistance to all drugs within two or more ARV drug classes. [NOTE: M184V/I is an exception and should not be considered when assessing this criterion. Prior HIV resistance testing is not required.]
* History of systemic corticosteroids (>14 days concurrent use), immunosuppressive anti-cancer or other immunosuppressive agents, interleukins, systemic interferons, systemic chemotherapy, or other medications considered significant by the investigator within the 24 weeks prior to study entry.
* ART initiated during acute infection (defined as p24, HIV NAAT, or HIV RNA PCR positive, and negative or indeterminate HIV antibody testing).
* Any history of receipt of therapeutic HIV vaccine or HIV monoclonal antibody therapy.
* Participation in any clinical study of an investigational product within 12 weeks prior to study entry or expected participation in such a study while on A5416.
* Known allergy/sensitivity or any hypersensitivity to components of either study agent or their formulation.
* Breastfeeding.
* Chronic hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg), hepatitis C antibody without documented history of prior treatment and clearance or virus RNA (HCV-RNA) or HCV antigen in blood at a Network-approved non-US laboratory that is EQA certified.
* Current untreated or incompletely treated active tuberculosis disease or untreated latent tuberculosis infection. [NOTE: Individuals who are on treatment for latent TB with at least 4 weeks of treatment completed are not excluded.]
* History of or current clinical atherosclerotic cardiovascular disease (ASCVD), as defined by 2013 American College of Cardiology/American Heart Association (ACC/AHA) guidelines, including a previous diagnosis of any of the following:

  * Acute myocardial infarction
  * Acute coronary syndromes
  * Stable or unstable angina
  * Coronary or other arterial revascularization
  * Stroke
  * Transient ischemic attack
  * Peripheral arterial disease presumed to be of atherosclerotic origin
* Diagnosis of cirrhosis.
* Diagnosis of untreated syphilis, gonorrhea, or chlamydia. [NOTE: Individuals who began treatment at least 3 days prior to study entry for any of the above are not excluded.]

No Step 2 and Step 3 Exclusion Criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a Grade ≥3 or higher systemic AE or any AE (regardless of grade) leading to premature study or treatment discontinuation | Step 1 Entry (Day 0) through to 48 weeks
  The proportion of participants reporting a Grade ≥3 systemic (i.e., not a local reaction) adverse event (AE) or any AE (regardless of grade) leading to premature study or treatment discontinuation at least possibly related (as judged by the CMC, blinded to active/placebo treatment) to the combination of 3BNC117-LS-J and 10-1074-LS-J.
  An AE is any unfavorable and unintended sign, symptom, or diagnosis occurring in a study participant during the conduct of the study regardless of the attribution. Adverse events are graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=potentially life-threatening, 5=death.
Viral suppression | Step 1 Entry (Day 0) through to Week 24
  The difference in proportion of participants with viral suppression during analytical treatment interruption (ATI) between those receiving 3BNC117-LS-J and 10-1074-LS-J and those receiving placebo. Viral suppression is defined as no confirmed HIV-1 RNA >200 copies/mL, at or prior to week 24 of ART discontinuation.

SECONDARY OUTCOMES:
Viral rebound at or prior to week 24 of ART discontinuation | Step 1 Entry (Day 0) through Week 24
  The cumulative probability of viral rebound at or prior to Week 24 in each treatment arm. Viral rebound is defined as confirmed HIV-1 RNA greater than 200 copies/mL.
HIV-1 RNA levels <50 copies/mL through week 24 of ART discontinuation | Step 1 Entry (Day 0) through Week 24
  The cumulative probability of participants maintaining HIV-1 RNA <50 copies/mL through Week 24 in each treatment arm.
Frequency of participants who do not meet the virologic or immunologic components of the ART resumption criteria while serum bNAb concentrations are ≥10 mcg/mL | Step 1 Entry (Day 0) until ART restart (Step 3 Entry)
  The number of participants in the active arm with serum bNAb concentrations (of both 3BNC-117-LS-J and 10-1074-LS-J) greater than or equal to 10 mcg/mL who have not met the viral load or CD4+ T cell components of the ART restart criteria at Step 1 and Step 2 study visits.
Frequency of participants who do not meet the virologic or immunologic components of the ART resumption criteria for 24 weeks after serum bNAb concentrations fall below 10 mcg/mL. | Step 1 Entry (Day 0) until ART restart (Step 3 Entry)
  The number of participants in the active arm with serum bNAb concentrations (of both 3BNC-117-LS-J and 10-1074-LS-J) less than 10 mcg/mL who have not met the viral load or CD4+ T cell components of the ART restart criteria at Step 1 and Step 2 study visits.
Frequency of participants who remain off ART and do not meet ART resumption criteria by study week in Step 1 and 2. | Step 1 Entry (Day 0) until ART restart (Step 3 Entry)
  The number of participants who remain of ART and do not meet ART resumption criteria will be tabulated at each study visit in Step 1 and 2.
Time to meeting the virologic or immunologic components of the ART resumption criteria. | Step 1 Entry (Day 0) until ART restart (Step 3 Entry)
  Time to meeting the viral load (virologic) or CD4+ T cell (immunologic) components of the ART resumption criteria estimated using Kaplan-Meier methods.
AUC of 3BNC117-LS-J and 10-1074-LS-J | Step 1 Entry (Day 0) through study follow-up
  The Area Under the Concentration (AUC) time curve for each participant calculated from available bNAb concentrations measured during study follow-up in the active treatment arm.
Clearance of 3BNC117-Ls-J and 10-1074-LS-J | Step 1 Entry (Day 0) until ART restart (Step 3 Entry)
  The clearance, describing the relationship between concentration and the rate of elimination from the body, for each participant will be calculated from available bNAb concentrations measured during study follow-up in the active treatment arm.
Concentration of 3BNC117-LS-J and 10-1074-LS-J at the time of viral rebound. | Step 1 Entry (Day 0) until ART restart (Step 3 Entry)
  The observed concentration of 3BNC117-LS-J and 10-1074-LS-J at the time of the first viral rebound (i.e., the first instance of confirmed HIV-1 RNA > 200 copies/mL) in the active treatment arm.
Number of participants who develop anti-3BNC117-LS-J and/or anti-10-1074-LS-J antibodies (ADA). | Step 1 Entry (Day 0) until ART restart (Step 3 Entry)
  The number of participants who develop anti-3BNC117-LS-J and/or anti-10-1074-LS-J antibodies at any point during study follow-up (cumulative incidence) in the active treatment arm.
CD4+ T-cell counts (cells/mm3) through entire study follow-up | Step 1 Entry (Day 0) through entire study follow-up
  Median CD4+ T-cell count at all required (i.e., not conditional) required visits during ATI and after ART restart in each treatment arm.
Percent of participants who develop anti-3BNC117-LS-J and/or anti-10-1074-LS-J antibodies (ADA). | Step 1 Entry (Day 0) until ART restart (Step 3 Entry)
  The percent of participants who develop anti-3BNC117-LS-J and/or anti-10-1074-LS-J antibodies at any point during study follow-up (cumulative incidence) in the active treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Mina Hosseinipour, MD, MPH, Study Chair — University of North Carolina Global HIV Prevention and Treatment CTU; Rebone Maboa, MBChB, DOHM, Study Chair — The Aurum Institute Pretoria CRS
Locations (9):
- Gaborone CRS (12701), Molepolole, Botswana
- Malawi (2):
  - Blantyre CRS (30301), Blantyre
  - Lilongwe Malawi CRS (12001), Lilongwe
- South Africa (6):
  - Ward 21 CRS (31966), Johannesburg, Gauteng
  - Soweto HVTN CRS (30351), Soweto, Gauteng
  - CAPRISA eThekwini CRS (31422), Durban, KwaZulu-Natal
  - Aurum Institute Klerksdorp CRS (30325), Klerksdorp, North West
  - Rustenburg CRS (31684), Rustenburg, North West
  - Groote Schuur HIV CRS (31708), Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/about-actg/templates-and-forms. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.

REFERENCES:
- See also: Related Info — https://actgnetwork.org